CLINICAL TRIAL: NCT05400005
Title: Impact of Different Types of Higher Dietary Protein Intake on Sleep Quality in Singapore Older Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Jung Eun Kim, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: S19
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Sleep; Gut Microbiome; Cardiometabolic Risk
Keywords: Dietary protein
MeSH Terms: interventions — Dietary Proteins

STUDY DESIGN:
Intervention Model Description: This is a 16-week factorial study design with subjects randomly assigned to consume normal-protein diet, higher-protein diet with micellar casein protein isolates or higher-protein diet with soy protein isolates. Subjects' sleep quality will also be evaluated and screened using the PSQI questionnaire (GSS ≤5 [good sleepers] vs. GSS >5 [poor sleepers]).
  Sixty-eight older men and women (aged 60-85y, approximately half men and half women) will be recruited with the expectation that ≥ 54 subjects (≥ 18 subjects per group) will complete the study (≤ 20% dropout rate). The 18 subjects recruited for each of the intervention group were further classified into poor (n=9) and good sleepers (n=9).
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Normal protein diet (control) (No Intervention): Subjects are to consume normal-protein diet based on the "My Healthy Plate" diet (launched by Health Promotion Board of Singapore) for the duration of the 16-week study.
- High protein diet (soy) (Experimental): Subjects are to consume higher-protein diet by following the "My Healthy Plate" diet (launched by Health Promotion Board of Singapore) and 20g of soy protein isolate for the duration of the 16-week study.
  Interventions: Other: Dietary protein
- High protein diet (Micellar Casein) (Experimental): Subjects are to consume higher-protein diet by following the "My Healthy Plate" diet (launched by Health Promotion Board of Singapore) and 20g of micellar casein isolate for the duration of the 16-week study.
  Interventions: Other: Dietary protein

INTERVENTIONS:
Other: Dietary protein — Intervention of the study include consuming a higher protein diet. Depending on the group allocation, this is done by asking the subjects to follow "My Healthy Plate" diet and consumption of 20g of protein isolates (casein or soy).
  Arms: High protein diet (Micellar Casein); High protein diet (soy)

SUMMARY:
Today, insufficient sleep has become a growing global problem. Sleep is essential to health and changes in sleep patterns are a part of the aging process. Inadequate and low-quality sleep also increases the risk for age-related cognitive decline and disease conditions. More importantly, due to COVID-19 health emergency, there is a significant increase of psychological distress and symptoms of mental illness and a worsening of quality of sleep. Therefore, there is an urgent need to investigate the way of improving sleep quality, in particular during and post COVID-19 period, in older adults.

One of the possible strategies in improving sleep quality with lifestyle modification is having higher-protein diet. However, this effect has not been fully elucidated in older adults. In addition, the effect of type of dietary protein on sleep quality is inconclusive and there is no clinical trial which assessed the differential response in sleep quality between animal-sourced protein vs. plant-sourced protein. Therefore, the purpose of this research project is to assess the impact of different types of higher dietary protein intake on sleep quality in Singapore older adults.

Findings from the proposed research will provide the scientific evidence of the beneficial effects of regularly consuming higher-protein diet on sleep quality in Singapore older adults. In addition, this research may validate the differential effect of different type of dietary protein on sleep quality. The results from the proposed research will also assist a practical guidance of nutritional behaviour changes providing sleep promoting effects to a large proportion of the Singapore population.

DETAILED DESCRIPTION:
During the 16-week intervention, subjects will be randomly assigned to 1 of 3 groups including consuming normal-protein diet, higher-protein diet supplemented with micellar casein protein or higher-protein diet supplemented with soy protein. Recommended Dietary Allowances for healthy Singaporean. Normal-protein diet will be designed following a healthy eating pattern diet, referred to as the "My Healthy Plate" launched by Health Promotion Board and subjects will consume 3 servings of dietary protein. Higher-protein diet will also follow a healthy eating pattern diet while subjects will additionally take either 20 g micellar casein protein isolate or 20 g soy protein isolate. One-on-one dietary counselling and written instructions for each subject will be provided by a research dietitian and trained research staff. Compliance with the diet interventions will be promoted by frequent online and in-person contact and dietary assessment. Blood amino acid concentration will also be assessed as an indicator of compliance to the protein intake.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 60-85 years old
2. Not following HPB diet

Exclusion Criteria:

1. Weight change > 3kg in the past 3 months
2. Exercise vigorously over the past 3 months
3. Drinking more than 2 alcoholic drinks per day
4. (if applicable) Pre-menopausal women
5. Taking dietary supplements or medications which may impact sleep outcomes (e.g. Nutritional Shakes (e.g. Ensure), Trp, 5-HTP or melatonin supplementations) the past 1 month
6. Taking dietary supplements which may impact the gut microbiota (e.g. antibiotics, prebiotics, probiotics) the past 2 months (a list of fermented foods)
7. Impaired renal function (normal values: estimated glomerular filtration rate ≥ 90 mL/min/1.73 m2 calculated by chronic kidney disease epidemiology collaboration equation; CKD EPI)
8. Soy intolerance and/or allergy or any medical conditions that may be affected by consumption of soy products (e.g. gout)
9. Prescribed and taking antihypertensive/cholesterol-lowering/ type-2 diabetic medication or Chinese medicine herb which started less than 3 years prior to the intervention participation
10. Diagnosed with gut/gastrointestinal issues such as lactose intolerance and irritable bowel syndrome (IBS)

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in sleep quality assessed by validated sleep questionnaires | Every 4 weeks (week 0, week 4, week 8, week 12 and week 16)
  Pittsburgh Sleep Quality Index Questionnaire (PSQI) will be used to assess the sleep quality. Overall score ranging from 0 to 21 points, where lower scores denote a healthier sleep quality.
Change in sleep quality assessed by electronic equipment | Every 4 weeks (week 0, week 4, week 8, week 12 and week 16)
  An electronic equipment, actigraphy, will be used to assess the sleep quality, including sleep timing and wake up timing.
Change in blood amino acid concentration | Every 8 weeks (week 0 , week 8 and week 16)
  Amino acid concentration in the blood will be measured
Change in blood serotonin concentration | Every 8 weeks (week 0 , week 8 and week 16)
  Serotonin concentration in the blood will be measured
Change in urinary 6-sulfatoxymelatonin (aMT6s) concentration | Every 8 weeks (week 0 , week 8 and week 16)
  6-sulfatoxymelatonin (aMT6s) concentration in the urine samples will be measured

SECONDARY OUTCOMES:
Change in fecal microbiome composition | Every 8 weeks (week 0 , week 8 and week 16)
  High-throughput sequencing method (using Illumina MiSeq platforms) will be used to assess the changes in gut microbiome composition
Change in fecal short chain fatty acid (SCFA) concentration | Every 8 weeks (week 0 , week 8 and week 16)
  SCFA concentration in fecal samples will be measured.
Change in serum lipopolysaccharide binding protein (LBP) concentration | Every 8 weeks (week 0 , week 8 and week 16)
  LBP concentration in blood samples will be measured.
Change in blood short chain fatty acid (SCFA) concentration | Every 8 weeks (week 0 , week 8 and week 16)
  SCFA concentration in the blood will be measured
Change in fecal bile acids | Every 8 weeks (week 0 , week 8 and week 16)
  Bile acids concentration will be determined from fecal samples of the subjects
Change in fecal zonulin | Every 8 weeks (week 0 , week 8 and week 16)
  Zonulin concentration will be determined from fecal samples of the subjects
Change in fecal calprotectin | Every 8 weeks (week 0 , week 8 and week 16)
  Calprotectin concentration will be determined from fecal samples of the subjects
Change in urinary creatinine concentration | Every 8 weeks (week 0 , week 8 and week 16)
  Creatinine concentration in the urine samples will be measured
Change in Estimated Glomerular Filtration Rate (eGFR) | Every 8 weeks (week 0 , week 8 and week 16)
  The estimated Glomerular Filtration Rate (eGFR) of the subjects will be measured from the blood
Change in Trimethylamine N-oxide (TMAO) | Every 8 weeks (week 0 , week 8 and week 16)
  Trimethylamine N-oxide (TMAO) concentration in the blood will be measured
Change in Blood Glucose | Every 8 weeks (week 0 , week 8 and week 16)
  Glucose concentration in the blood will be measured
Change in Blood Triglyceride | Every 8 weeks (week 0 , week 8 and week 16)
  Triglyceride concentration in the blood will be measured
Change in Blood Cholesterol | Every 8 weeks (week 0 , week 8 and week 16)
  Total cholesterol concentration in the blood will be measured
Change in Blood Low-density Lipoprotein-cholesterol (LDL) | Every 8 weeks (week 0 , week 8 and week 16)
  LDL concentration in the blood will be measured
Change in Blood High-density Lipoprotein-cholesterol (LDL) | Every 8 weeks (week 0 , week 8 and week 16)
  HDL concentration in the blood will be measured
Change in Blood Advanced Glycation End-product (AGEs) | Every 8 weeks (week 0 , week 8 and week 16)
  AGEs concentration in the blood will be measured
Change in Skin Advanced Glycation End-product (AGEs) | Every 8 weeks (week 0 , week 8 and week 16)
  Using a scanner, the AGEs levels in the skin will be measured
Change in Blood Interleukin-6 (IL-6) | Every 8 weeks (week 0 , week 8 and week 16)
  Interleukin-6 (IL-6) concentration in the blood will be measured
Change in Endothelial Function | Baseline and Post-intervention (week 0 and week 16)
  Endothelial functions are determined by the function of endothelial progenitor cells
Change in Flow Mediate Dilation | Baseline and Post-intervention (week 0 and week 16)
  Flow mediate dilation (%)
Change in weight and height | Every 4 weeks (week 0, week 4, week 8, week 12 and week 16)
  Weight (in kilograms) and height (in meters) will be combined to report BMI in kg/m^2
Change in waist circumference | Every 4 weeks (week 0, week 4, week 8, week 12 and week 16)
  Waist circumference (in cm) will be measured
Change in blood pressure | Every 4 weeks (week 0, week 4, week 8, week 12 and week 16)
  Systolic and diastolic blood pressure (in mmHg) will be measured by a blood pressure monitor.
Dietary assessment | Every 4 weeks (week 0, week 4, week 8, week 12 and week 16)
  Dietary assessment will be assessed by 3-day dietary food record
Change in mood (stress) | Every 4 weeks (week 0, week 4, week 8, week 12 and week 16)
  Perceived Stress Scale (PSS) will be used to assess the stress levels
Change in mood (depression) | Every 4 weeks (week 0, week 4, week 8, week 12 and week 16)
  Geriatric Depression Scale (GDS) Assessment will be used to assess the depression status
Change in mood (anxiety) | Every 4 weeks (week 0, week 4, week 8, week 12 and week 16)
  Geriatric Anxiety Inventory (GAI) Assessment will be used to assess the anxiety status.

CONTACTS AND LOCATIONS:
Overall Officials: Jung Eun Kim, PhD, Principal Investigator — National University of Singapore
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Electronic copies of the data with identifiable participant information will be kept on a secure website with access limited to Dr. Kim and her research staff. All data will be de-identified prior to statistical analyses.

REFERENCES:
- [Background] Cappuccio FP, D'Elia L, Strazzullo P, Miller MA. Sleep duration and all-cause mortality: a systematic review and meta-analysis of prospective studies. Sleep. 2010 May;33(5):585-92. doi: 10.1093/sleep/33.5.585. PMID 20469800
- [Background] Sutanto CN, Wang MX, Tan D, Kim JE. Association of Sleep Quality and Macronutrient Distribution: A Systematic Review and Meta-Regression. Nutrients. 2020 Jan 2;12(1):126. doi: 10.3390/nu12010126. PMID 31906452
- [Background] Zhou J, Kim JE, Armstrong CL, Chen N, Campbell WW. Higher-protein diets improve indexes of sleep in energy-restricted overweight and obese adults: results from 2 randomized controlled trials. Am J Clin Nutr. 2016 Mar;103(3):766-74. doi: 10.3945/ajcn.115.124669. Epub 2016 Feb 10. PMID 26864362
- [Background] Rosenfield AT, Zeman RK, Cronan JJ, Kay CJ. Ultrasound in the evaluation of renal masses. Conn Med. 1980 Jan;44(1):1-5. No abstract available. PMID 7353359
- [Background] St-Onge MP, Crawford A, Aggarwal B. Plant-based diets: Reducing cardiovascular risk by improving sleep quality? Curr Sleep Med Rep. 2018 Mar;4(1):74-78. Epub 2018 Feb 5. PMID 29910998
- [Derived] Yao Y, Mak IE, Sutanto CN, Leong ZN, He Q, Pahwa U, Ling LH, Khoo CM, Ackers-Johnson MA, Foo RS, Kim JE. Impact of quantity and source of dietary protein intake within a healthy dietary pattern on cardiovascular disease risk factors in Singapore older adults: a randomized controlled trial. Food Funct. 2025 Dec 8;16(24):9533-9544. doi: 10.1039/d5fo03817k. PMID 41284351